CLINICAL TRIAL: NCT07284758
Title: A Phase 2, Open-Label, Single-Arm, Multicenter Study to Evaluate the Efficacy of Cemsidomide + Dexamethasone in Subjects With Relapsed/Refractory Multiple Myeloma
Brief Title: A Study to Evaluate the Efficacy of Cemsidomide + Dexamethasone in Participants With Relapsed/Refractory Multiple Myeloma
Acronym: MOMENTUM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: C4 Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFT7455-2101
Record Dates: First submitted 2025-12-09; First posted 2025-12-16 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma; Relapsed/Refractory Multiple Myeloma
Keywords: cemsidomide; dexamethasone; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cemsidomide + Dexamethasone: (Experimental): Participants receive cemsidomide plus dexamethasone during a 28-day treatment cycle, and will continue to receive treatment until the participant meets one of the discontinuation criteria.
  Interventions: Drug: Cemsidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Cemsidomide — dosed orally (PO) once a day (QD) 14 days on/14 days off for each 28-day cycle
Drug: Dexamethasone — dosed PO once a week (QW) on Days 1, 8, 15, and 22 for each 28-day cycle

SUMMARY:
This is a Phase 2, open-label, single-arm, multicenter study to assess the antimyeloma activity and further characterize the safety, tolerability, PK, and PD of cemsidomide in combination with dexamethasone in participants with relapsed/refractory multiple myeloma (r/r MM).

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide signed informed consent for the study.
2. Age ≥ 18 years at the time of signed consent.
3. Subjects must have a documented diagnosis of MM and measurable disease at enrollment.
4. Received at least 3 prior anti-myeloma regimens (for a minimum of 2 or more consecutive cycles) that must have included an immunomodulatory drug (i.e., IKZF 1/3 degrader), a proteasome inhibitor, an anti-CD38 antibody, and a T-cell engager (TCE) or chimeric antigen receptor T-cell (CAR-T) therapy, unless not available per local standard of care.
5. Subjects need to have adequate organ function.
6. Toxicities from prior anticancer therapies must have resolved to baseline severity or CTCAE ≤ Grade 1.
7. Female subjects may not be pregnant or intend to become pregnant, may not breastfeed or intend to breastfeed, or donate ova during their participation in this study until 30 days after the last dose of study treatment.
8. Male subjects must agree to use a condom when having intercourse with a person of childbearing potential during the Treatment Period and for at least 30 days after the last dose of study treatment.
9. Male subjects must refrain from donating sperm during the Treatment Period and for 30 days after discontinuation.
10. Subjects must refrain from donating blood during study treatment and for 30 days after discontinuation.

Exclusion Criteria:

1. Presence of myeloma in the central nervous system (CNS).
2. Subjects with any of the following:

   * Systemic light chain amyloidosis
   * Polyneuropathy, Organomegaly, Endocrinopathy, Monoclonal gammopathy, and Skin changes (POEMS) Syndrome
   * Myelodysplastic syndrome (MDS).
3. Previously treated with cemsidomide.
4. Clinically significant impaired cardiac function or cardiac disease.
5. Thromboembolic event within 3 months prior to enrollment.
6. Known malignancy other than study indication that has progressed or required treatment within the past 3 years.
7. Uncontrolled active bacterial, fungal, or viral infection.
8. Inability or difficulty swallowing tablets.

NOTE: Other inclusion/exclusion criteria may apply, per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) per International Myeloma Working Group (IMWG) Response Criteria by an Independent Review Committee (IRC) | up to approximately 43 months

SECONDARY OUTCOMES:
Duration of response (DoR; IRC assessed) | up to approximately 43 months
Complete response (CR) rate (IRC assessed) | up to approximately 43 months
Time to response (IRC assessed) | up to approximately 43 months
Progression free survival (PFS; IRC assessed) | up to approximately 43 months
Overall survival (OS) | up to approximately 43 months
Adverse events (AEs); serious AEs (SAEs); AEs leading to treatment interruption, reduction, or discontinuation; and deaths | within 30 to 35 days of the last dose of study treatment
Plasma concentrations of cemsidomide | up to approximately 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Binod Dhakal, M.D., Principal Investigator — Medical College of Wisconsin; Martin Kaiser, M.D., Principal Investigator — The Royal Marsden; Aurore Perrot, M.D., Principal Investigator — Universite de Toulouse
Locations (1):
- Berenson Cancer Center, West Hollywood, California, United States

IPD SHARING:
Plan to Share IPD: No